CLINICAL TRIAL: NCT04463953
Title: A Phase 2 Clinical Trial to Evaluate the Efficacy of Zanubrutinib Plus Ixazomib and Dexamethasone in Newly Diagnosed Symptomatic Waldenström Macroglobulinemia
Brief Title: Zanubrutinib, Ixazomib and Dexamethasone in Patients With Treatment Naive Waldenstrom's Macroglobulinemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2020002
Record Dates: First submitted 2020-07-04; First posted 2020-07-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2024-05

CONDITIONS: Waldenström Macroglobulinemia
Keywords: Waldenström Macroglobulinemia; Zanubrutinib; Ixazomib; Dexamethasone
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — zanubrutinib; ixazomib; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Zanubrutinib, 160mg orally, twice a day; Ixazomib, 4 mg orally, day 1, 8, 15; Dexamethasone, 20mg orally, days 1, 8, 15.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ZID regimen (Experimental): Zanubrutinib, 160mg orally, twice a day; Ixazomib, 4 mg orally, day 1, 8, 15; Dexamethasone, 20mg orally, days 1, 8, 15.
  Interventions: Drug: Zanubrutinib,Ixazomib and Dexamethasone

INTERVENTIONS:
Drug: Zanubrutinib,Ixazomib and Dexamethasone — Zanubrutinib, 160mg orally, twice a day; Ixazomib, 4 mg orally, day 1, 8, 15; Dexamethasone, 20mg orally, days 1, 8, 15；Ixazomib and dexamethasone every 4 weeks of a cycle, with induction of 6 cycles, and then maintain every 12 weeks, up to 6 cycles (96 cycles in total). Zanubrutinib is taken orally twice a day for up to 96 cycles, with a reduction in the last ID cycle. ZID regimen will continue 6 cycles after reaching the maximum response after introduction section.

SUMMARY:
This study aims to evaluate the efficacy of BTK inhibitor Zanubrutinib combined with Ixazomib and Dexamethasone (ZID) for the newly diagnosed Waldenstrom Macroglobulinemia. This ZID regimen will be given up to 24 months and stopped for observation. We propose this combination will improve the deep remission (≥VGPR) compared to single Zanubrutinib or IRD regimen and can be a time-limited regimen which will reduce the life-time therapy and benefit the patients.

DETAILED DESCRIPTION:
As Waldenstrom Macroglobulinemia cells always have two or three components tumor cells, including lymphocyte, Lymphoplasmacytic cells and plasma cells. We designed a oral regimen to target both lymphoma cells (Zanubrutinib) and plasma cells (Ixazomib plus Dexamethasone) to eliminate the tumor cells of WM. We propose this combination will improve the deep remission of WM (≥VGPR) . Zanubrutinib will be given 160mg Bid per day, up to 24 months, Ixazomib 4mg per week and Dexamethasone 20mg per week for three weeks, every 4 weeks one course. ID will be given 6 course as introduction and then one course every 12 weeks for up to 24 months. At the last ID course, Zanubrutinib will be stopped. The last ID course is to prevent the bounce of IgM because of Zanubrutinib discontinue.

ELIGIBILITY:
Inclusion Criteria:

1. The gender of the patient is not limited, and the age is ≥18 years old;
2. Must meet WM's diagnostic standards;
3. The patient is an untreated or patient who has not undergone standard treatment. The specific conditions are as follows:

   1. No combined chemotherapy with BR, RCD, VRD, CHOP and COP
   2. No treatment regimen containing fludarabine
   3. Chlorambucil or cyclophosphamide for less than 4 weeks (alone or in combination with adrenal glucocorticoids)
   4. The above treatment did not reach the treatment response (MR)
   5. If the above treatment has been applied, the treatment needs to be stopped for 2 weeks before entering the group to start treatment
4. The indications for the treatment of indolent lymphoma mainly include (at least one of the following conditions):

   1. Symptomatic hyperviscosity;
   2. symptomatic peripheral neuropathy;
   3. Amyloidosis;
   4. Cold agglutinin disease; cryoglobulinemia;
   5. Disease-related cytopenia (Hb<100 g/L, PLT<100×10^9/L);
   6. giant lymph nodes;
   7. Those with systemic systemic symptoms: for two weeks/recurrent fever (above 38℃) and not caused by infection, or Night sweats and/or weight loss >10% within 6 months;
   8. The disease progresses rapidly, for example, the lymph nodes increase by more than 50% within 2 months, and/or peripheral blood lymphocytes absolute value doubling time <6 months, and/or rapid hemoglobin or platelet non-autoimmune causes slow down
   9. When there is evidence that the disease has transformed.
5. ECOG score ≤ 2 points
6. Laboratory examination: neutrophils ≥ 0.75×10^9/L; platelets ≥ 50×10^9/L; total bilirubin ≤ 2.5 times upper limit; alanine aminotransferase/aspartate aminotransferase ≤3 times upper limit. Creatinine clearance rate ≥ 30ml/min.
7. The patient's expected survival time is ≥ 3 months.

Exclusion Criteria:

1. Malignant tumors (including active central nervous system lymphoma) other than B-NHL have been diagnosed or treated within the past year;
2. There is clinical evidence that large cell lymphoma transformation has occurred;
3. Non-lymphoma-related liver and kidney damage: alanine aminotransferase (ALT)> 3 times the upper limit of normal value, aspartate aminotransferase (AST)> 3 times the upper limit of normal value, total bilirubin (TBIL)> upper limit of normal value 2 Times, serum creatinine clearance rate <30ml/min;
4. Other serious medical conditions will affect the study (such as uncontrolled diabetes, gastric ulcers, other serious cardiopulmonary diseases, etc.). The decision-making power belongs to the researcher;
5. Known history of infection with human immunodeficiency virus (HIV) or active hepatitis B virus (HBV) infection, or any uncontrolled active systemic infection requiring intravenous antibiotics.
6. Central nervous system dysfunction with clinical manifestations or central invasion (Bing-Neel syndrome);
7. Patients who have undergone major surgery (not including lymph node biopsy) within the past 14 days or expected major surgery during treatment;
8. Inability to swallow capsules or suffer from malabsorption syndrome, diseases that significantly affect gastrointestinal function, have undergone gastric or small bowel resection, symptomatic inflammatory bowel disease or ulcerative colitis, partial or complete intestinal obstruction.
9. Need to receive strong cytochrome P450 (CYP) 3A inhibitor treatment.
10. Women who are pregnant or breastfeeding, women of childbearing age who have not taken contraception;
11. Allergy to the drugs used.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Deep remission response rate | up to 5 years
  ≥VGPR after 6 cycles introduction

SECONDARY OUTCOMES:
Complete response (CR) | up to 12 months
  Disappearance of monoclonal protein on immunofixation (both serum and urine); No histologic evidence of bone marrow involvement; Resolution of adenopathy and/or organomegaly on CT; Resolution of clinical signs or symptoms attributed to WM/LPL.
Progress-free survival (PFS) | up to 5 years
  the time from treatment initiation until disease progression or death
Duration of response (DoR) | up to 5 years
  the time from best response (R) to progression/death (P/D)
Overall survival (OS) | up to 36 months
  The percentage of patients in treatment group who are still alive for a certain period of time after they were diagnosed with Waldenstrom's Macroglobulinemia.
Time to next treatment (TTNT) | up to 5 years
  time from end of primary treatment to institution of next therapy
Overall response | up to 5 year
  minimor response+partial response+VGPR+CR

CONTACTS AND LOCATIONS:
Overall Officials: Shuhua Yi, Principal Investigator — Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Treon SP, Xu L, Guerrera ML, Jimenez C, Hunter ZR, Liu X, Demos M, Gustine J, Chan G, Munshi M, Tsakmaklis N, Chen JG, Kofides A, Sklavenitis-Pistofidis R, Bustoros M, Keezer A, Meid K, Patterson CJ, Sacco A, Roccaro A, Branagan AR, Yang G, Ghobrial IM, Castillo JJ. Genomic Landscape of Waldenstrom Macroglobulinemia and Its Impact on Treatment Strategies. J Clin Oncol. 2020 Apr 10;38(11):1198-1208. doi: 10.1200/JCO.19.02314. Epub 2020 Feb 21. PMID 32083995
- [Background] Treon SP, Xu L, Hunter Z. MYD88 Mutations and Response to Ibrutinib in Waldenstrom's Macroglobulinemia. N Engl J Med. 2015 Aug 6;373(6):584-6. doi: 10.1056/NEJMc1506192. No abstract available. PMID 26244327
- [Background] Castillo JJ, Meid K, Gustine JN, Dubeau T, Severns P, Hunter ZR, Yang G, Xu L, Treon SP. Prospective Clinical Trial of Ixazomib, Dexamethasone, and Rituximab as Primary Therapy in Waldenstrom Macroglobulinemia. Clin Cancer Res. 2018 Jul 15;24(14):3247-3252. doi: 10.1158/1078-0432.CCR-18-0152. Epub 2018 Apr 16. PMID 29661775